CLINICAL TRIAL: NCT02666534
Title: A Randomised Trial Comparing Methyl Aminolaevulinate Photodynamic Therapy With and Without Ablative Fractional Laser Treatment in Patients With Microinvasive Squamous Cell Carcinoma: Results From a 24-month Follow-up
Brief Title: Efficacy of AFL-assisted PDT in Microinvasive Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Song Ki-Hoon, Associate professor, Dong-A University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DAUderma-05
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Microinvasive Squamous Cell Carcinoma
Keywords: Ablative fractional laser; microinvasive squamous cell carcinoma; photodynamic therapy
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AFL-PDT (Experimental): Forty-five Korean patients were enrolled in this study. Patients were randomly assigned to receive either AFL-PDT or MAL-PDT in a 1:1 ratio. As result, the patients were randomized to treatment with AFL-PDT (21 patients) or MAL-PDT (24 patients)
  Interventions: Drug: lidocaine-prilocaine 5% cream application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: methyl-aminolevulinate application; Device: Illuminating using red light-emitting diode lamps
- MAL-PDT (Active Comparator): Forty-five Korean patients were enrolled in this study. Patients were randomly assigned to receive either AFL-PDT or MAL-PDT in a 1:1 ratio. As result, the patients were randomized to treatment with AFL-PDT (21 patients) or MAL-PDT (24 patients)
  Interventions: Drug: methyl-aminolevulinate application; Device: Illuminating using red light-emitting diode lamps

INTERVENTIONS:
Drug: lidocaine-prilocaine 5% cream application — The lesions were then cleansed with saline gauze, and a lidocaine-prilocaine 5% cream (EMLA®; Astra Pharmaceuticals, LP, Westborough, MA, USA) was applied to the treatment area for 30 min under occlusion
  Arms: AFL-PDT
Device: 2940-nm Er:YAG AFL pretreatment — After the anesthetic cream was removed, AFL was performed using a 2940-nm Er:YAG AFL (Joule; Sciton, Inc., Palo Alto, CA, USA) with a 500 µm ablation depth, level 1 coagulation, 22% treatment density, and a single pulse
  Arms: AFL-PDT
Drug: methyl-aminolevulinate application — Immediately after the AFL, a 1-mm thick layer of methyl-aminolevulinate (16% Metvix® cream; PhotoCure ASA, Oslo, Norway) was applied to the lesion and to 5 mm of the surrounding healthy tissue. The area was covered with an occlusive dressing (Tegaderm; 3M, Co., Saint Paul, MN, USA) for 3 h, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's light.
Device: Illuminating using red light-emitting diode lamps — Each treatment area was then separately illuminated using red light-emitting diode lamps (Aktilite CL128; Galderma S.A., Bruchsal, Germany) with peak emission at 632 nm and a total light dose of 37 J/cm2. Areas scheduled to receive MAL-PDT received the second treatment 7 days later. During the illumination, patients were asked to evaluate pain intensity using an 11-point visual analog scale.

SUMMARY:
Surgical excision is the standard treatment for cutaneous SCC. However, many patients diagnosed with SCC are elderly and ineligible for surgery. Ablative fractional laser- assisted photodynamic therapy (AFL-PDT) offered a higher efficacy than conventional Methylaminolevulinate (MAL)-PDT.

DETAILED DESCRIPTION:
Squamous cell carcinoma (SCC) lesions are potentially metastatic and can be life threatening. Hence, surgical excision is the standard treatment for cutaneous SCC. However, some patients are ineligible for surgery because of their poor general health, concomitant anticoagulant or immunosuppressive therapies, or allergy to local anesthetics.

Photodynamic therapy (PDT) with methylaminolevulinate (MAL) is an innovative treatment modality that has been approved in Europe for the treatment of actinic keratosis, basal cell carcinoma, and Bowen's disease. However, currently, there is insufficient evidence to support the routine use of topical PDT for SCC.

Ablative fractional laser (AFL) ablates the epidermis and dermis without significant thermal injury, creating microscopic ablation zones in the portion of the skin that the laser is applied to. Our previous studies showed that AFL-primed MAL-PDT (AFL-PDT) offered a higher efficacy than conventional MAL-PDT in the treatment of many other diseases, such as actinic keratosis, actinic cheilitis, and Bowen's disease.

Investigators recruited Korean patients with microinvasive SCC and compared the efficacy, recurrence rate, and cosmetic outcomes of AFL-PDT with those of standard MAL-PDT.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more who had previously untreated microinvasive SCC, providing they satisfied both of the following conditions:

  * tumor invasion into the papillary dermis (Clark level II) according to a biopsy specimen and
  * difficulty in surgical excision because of health problems (bleeding tendency or cardiac problems)

Exclusion Criteria:

* pregnancy or lactation
* active systemic infectious disease
* other inflammatory, infectious, or neoplastic skin diseases in the treated area
* allergy to MAL,other topical photosensitizers, or excipients of the cream
* history of photosensitivity
* use of immunosuppressive or photosensitizing drugs
* participation in any other investigational study in the preceding 30 days
* history or indicators of poor compliance
* Histological findings of acantholysis, desmoplasia, perineural or lymphovascular invasion, and echographic features of regional lymph node metastasis were the disease-specific exclusion criteria

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Difference of short-term complete response (CR) rate between AFL-PDT and MAL-PDT | Short-term CR rate was evaluated at 3 months
  The response was classified as either complete response (complete disappearance of the lesion) or incomplete response (incomplete disappearance of the lesion)
Difference of long-term complete response (CR) rate between AFL-PDT and MAL-PDT | Long-term CR rate was evaluated at 24 months
  The response was classified as either complete response (complete disappearance of the lesion) or incomplete response (incomplete disappearance of the lesion)
Difference of recurrence rate at 24 months | Recurrent rate was evaluated at 24months
  In all cases of complete response, the patients were reviewed at 24 months to check for recurrence. Post-therapy punch biopsies were performed when there was doubt concerning incomplete-response and clinical recurrence

SECONDARY OUTCOMES:
Difference of the cosmetic outcome between AFL-PDT and MAL-PDT | Cosmetic outcome was assessed by each investigator for all lesions that achieved a complete response at 24 months
  The overall cosmetic outcome was assessed by each investigator for all lesions that achieved complete response at 24 months, and was graded using a 4-point scale: excellent (only slight occurrence of redness or change in pigmentation), good (moderate redness or change in pigmentation), fair (slight to moderate scarring, atrophy, or induration), or poor (extensive scarring, atrophy, or induration)

OTHER OUTCOMES:
Differences of Adverse events(erythema, burning sensation, swelling, bleeding) between AFL-PDT and MAL-PDT | Within 24 months after each treatment
  Adverse events reported by the patients were noted at each follow-up visit, including severity, duration, and need for additional therapy. All events due to PDT were described as phototoxic reactions(e.g erythema, burning sensation, swelling, bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-A University, Busan, Dong Dae Sin-dong, Seo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi SH, Kim KH, Song KH. Effect of Methyl Aminolevulinate Photodynamic Therapy With and Without Ablative Fractional Laser Treatment in Patients With Microinvasive Squamous Cell Carcinoma: A Randomized Clinical Trial. JAMA Dermatol. 2017 Mar 1;153(3):289-295. doi: 10.1001/jamadermatol.2016.4463. PMID 28199463